CLINICAL TRIAL: NCT01867502
Title: A 12-week Study to Compare the Effects of Vildagliptin Versus Glibenclamide on Glycemic Variability After a Sub Maximal Exercise Test in Patients With Type 2 Diabetes Inadequately Controlled With Metformin.
Brief Title: Effects of Vildagliptin Versus Glibenclamide on Glycemia After Exercise in Patients With Type 2 Diabetes
Acronym: DIABEX-VILDA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237ABR05T; 12-0444 (Other: Research Group and Post Graduation)
Record Dates: First submitted 2013-05-17; First posted 2013-06-04 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2; Hypoglycemic Agents; Diabetic Blood Glucose Monitoring; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Vildagliptin; Glyburide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MET + Glibenclamide Group (Other): Usual Metformin stipulated: 500 or 850mg 3 times a day, if tolerated by patients.
  The initial dose of glibenclamide group will be 5mg / day during the first week of study, later it will increase to 10 mg / day (2 x 5mg). When the adjustments will be done, the dose may reaching the maximum dose allowed, which is 20 mg / day.
  Interventions: Drug: MET + Glibenclamide Group
- MET + Vildagliptin Group (Other): Usual Metformin stipulated: 500 or 850mg 3 times a day, if tolerated by patients.
  Vidagliptin group will receive 50mg of this drug twice a day during 12 weeks.
  Interventions: Drug: MET + Vildagliptin Group

INTERVENTIONS:
Drug: MET + Vildagliptin Group — Vidagliptin group will receive 50mg of this drug twice a day during 12 weeks added to usual metformin.
  For the glicemic control evaluation will be used the capilar glycemia at home. The adjustments will be done by the researcher coordinator.
  Other Names: Galvus®; Glyburide; Glucophage
  Arms: MET + Vildagliptin Group
Drug: MET + Glibenclamide Group — The initial dose of glibenclamide group will be 5mg / day during the first week of study, later it will increase to 10 mg / day (2 x 5mg). With the control the dose may be adjusted, reaching the maximum dose allowed, which is 20 mg / day.
  For the glycemic control evaluation will be used the capillar glycemia at home. The adjustments will be done by the researcher coordinator.
  Other Names: Daonil®; Glucophage
  Arms: MET + Glibenclamide Group

SUMMARY:
Exercise is considered a way to benefit the health of unhealthy and healthy individuals. This is confirmed by different scientific researches, in which people who participated improve their health. The present study will be conducted to test the hypothesis that vildagliptin associated with metformin may have more impact in improving glucose variability after a sub-maximal exercise test, as compared to glibenclamide. Our general aim will be to evaluate glucose variability after the submaximal exercise test under the treatment with vildagliptin or glibenclamide. The specific aims of this study are to evaluate the oxidative stress, endothelial function, metabolic and cardiovascular responses to exercise under the treatment with vildagliptin or glibenclamide. All these responses are important in patients with Diabetes Mellitus type II. Allied to the patient's routine treatment (metformin), they will receive orally a second drug, to take in 12 weeks. The patients will be raffled to take one of the two drugs that act on glycemia, that are called vildagliptin (50 mg of this drug twice a day) and glibenclamide (5 mg once a day during the first week and later you will increase to 5 mg twice a day). The metformin drug will continue be used.

Patients who meet the eligible criteria for the study will first make the test of the maximum effort, to determination of peak oxygen consumption (VO2peak) and ventilatory thresholds. Forty eight hours after this test, patients will be allowed to do the pre-drugs protocol that will be given in three consecutive days as explained below.

* Day 1: Begin a 24-hour urinary collection, perform vascular doppler ultrasound to evaluate endothelial function and then the glucose sensor will be inserted subcutaneously (begin continuous glucose monitoring system - CGMS evaluation);
* Day 2: End the 24-hour urinary collection, submit to the submaximal test (blood collection at baseline, 15 and 30 min of the session, and 60 min after recovery). On the same day, the patients will begin 24h ambulatory blood pressure monitoring (24h-ABPM).
* Day 3: Removal of the glucose sensor; end of the 24h ABPM, randomization. This same protocol, except the randomization will be repeated at the end of the 12 week treatment.

DETAILED DESCRIPTION:
The main procedures will occur during three consecutive days, before randomization and 3 days before 12 weeks. In the first day, the patients will begin the 24hour urinary collection; the ultrasonography will be made in fasting state and they will place the sensors (CGMS and MAPA). In the second day, the blood samples will be collected and the patients will undergo sub-maximal exercise test; in the third day the sensors will be removed. The sub-maximal exercise test will occur on day 2 after a standard breakfast (500 kcal; 60% carbohydrate, 30% fat and 10% protein) after 8 hours overnight fast. After the three days of the first assessments, the selected patients will be divided into two groups, the group 1 receiving vildagliptin and the group 2 receiving glibenclamide for 12 weeks. There will be follow up visits on week 4 and 8. The variables in response to exercise (sub-maximal test) will be compared between the groups after 12 weeks.

The sample estimated will be 20 patients (10% drop out included) with DM2, from outpatient clinics of Serviço de Endocrinologia do Hospital de Clínicas de Porto Alegre (HCPA) or from public health. Patients will be randomized to metformin plus vildagliptin (MET + vilda), which will receive an additional vidagliptin dose of 50 mg twice a day and metformin plus glibenclamide group (MET + gliben) that will receive an additional glibenclamide dose of 5 - 20 mg once a day. Based on Marfella et al (13) study on the evaluation of the efficacy of treatment with Vildagliptin or Sitagliptin on blood glucose in patients with DM2 inadequately controlled with Metformin, a sample size with a 90% power and one alpha (α) of 0, 01 was calculated. Vidagliptin had a serious effect (51% reduction in MAGE), since the average difference was 25mg/dl with a 16 and 7mg/dl SD. After 20 subjects were analyzed, the calculated sample will be redone for confirming the sample efficacy for evidence of the expected effect evidence.

Adverse events, including serious adverse events or pregnancies will be collected and reported in the medical report of the study (Annex IV).

The reports containing serious adverse events or pregnancies will be forwarded to the respective manufacturer laboratory within 24 hrs after their knowledge, and the health authority according to the local law.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (fasting glucose ≥ 126 mg/dl or 7.0 mmol/l)(25);
* Recent HbA1C determination (between 7, 5 and 10%);
* Not involved in regular physical exercise;
* Older than 18 years;
* In use of Metformin.

Exclusion Criteria:

* Smoker and use of analgesic or anti-inflammatory drugs during the week of the study
* BMI > 40 kg/m²;
* Proliferative retinopathy;
* Ischemic cardiomyopathy;
* Peripheral vascular disease;
* Blood Aspartate transaminase (AST) and Alanine transaminase (ALT) 2.5 times higher the normal concentration before screening visit
* Lactose intolerance;
* Renal insufficiency (creatinine clearance <60ml/min);
* Blood pressure more than 180/100mmHg at rest (3 consecutive measures).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Change in Glycemic variability | Baseline and 12 weeks
  Continuous glucose monitoring system (CGMS) during 48 hours (24h before and 24 after the submaximal exercise test).

SECONDARY OUTCOMES:
Change in Hemodynamic response to exercise: Cardiac output (Q), Stroke Volume (SV) and blood pressure (BP) | Each 2 minutes during exercise and until 60 min post in baseline and 12 weeks
  Cardiac output (Q) and the Stroke Volume (SV)and blood pressure (BP) will be measured before the sub-maximal tests, 10% below the second threshold and every 2 minutes of recovery.

OTHER OUTCOMES:
Change in Flow Mediated Dilatation (FMD) | Baseline and 12 weeks
  This analysis will be performed by a high-resolution ultrasound of the brachial artery (doppler vascular), which characterizes the Flow Mediated Dilatation (FMD), which is expressed by changes in basal diameter in response to the increased flow and Nitroglycerin (NTG), which will be applied in a single dose (0.4 mg) as a sublingual spray.
Change in Blood pressure variability | Baseline and 12 weeks
  Blood Pressure Monitoring Sensor (BPMS)which will be programmed to automatically measuring the blood pressure every 15 minutes during the day (06:00 to 22:00 h), and every 20 minutes during the night (22:00 to 6:00 h.
Change in Plasma glucagon concentration on exercise | -1h, 0, 15min, 30 min (end), 60min post exercise in baseline and 12 weeks
  EDTA Vacutainer tubes of 10 ml will be used to perform the blood tests and they will be stored at -20º to send them to the Molecular and Proteins Analysis Unit after buying specific kit.
Change in Oxidative stress (F2 isoprostane 8-iso prostaglandin F2α); | Baseline and 12 weeks.
  The 24-hour urinary samples will be collected at visit 1 and 4 to evaluate the oxidative stress. Free 8-iso PGF2α that is most frequently measured F2 isoprostane in body fluids.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz BS Schaan, PhD, Principal Investigator — Federal University of Rio Grande do Sul; Aline AF Fofonka, MSc, Study Chair — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Fofonka A, Ribeiro JP, Casali KR, Schaan BD. Effects of vildagliptin compared with glibenclamide on glucose variability after a submaximal exercise test in patients with type 2 diabetes: study protocol for a randomized controlled trial, DIABEX VILDA. Trials. 2014 Nov 4;15:424. doi: 10.1186/1745-6215-15-424. PMID 25366037